CLINICAL TRIAL: NCT03444311
Title: Development of Combined Nutritional Therapies for the Treatment of Ulcerative Colitis Through the Increase of the Biodiversity of the Microbiota.
Brief Title: Combined Nutritional Therapies for the Treatment of Ulcerative Colitis
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Low tolerability of fibers included in the product
Sponsor: AB Biotics, SA (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RETOS
Record Dates: First submitted 2018-02-08; First posted 2018-02-23 (Actual); Last update posted 2020-07-08 (Actual); Status verified 2020-07

CONDITIONS: Colitis, Ulcerative
Keywords: microbiota; ulcerative colitis; fiber; probiotic
MeSH Terms: conditions — Colitis, Ulcerative

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- A: 1 dosis (Active Comparator): 1 dosis (3E+09 cfu/day + 6 g of fiber/day)
  Interventions: Dietary Supplement: A: 1 dosis
- B: 2 dosis (Active Comparator): 2 dosis (3E+09 cfu/day + 12 g of fiber/day)
  Interventions: Dietary Supplement: B: 2 dosis

INTERVENTIONS:
Dietary Supplement: A: 1 dosis — 1 dosis (3E+09 cfu/d + 6 g of fiber) Two different combinations of fibers (formula A and B) will be tested with the following administration pattern for both groups.
  Week 1: Formula A Week 2: Formula A Week 3: Formula B Week 4: Formula B
  Composition of an envelope of formula A:
  Formula A Composition (g) Pectin 1 B-glucan oatmeal 0.25 High-grade polymerization inulin 1.75 Inulin of low degree of polymerization 1,5 Polydextrose 1 Guar gum partially hydrolyzed 0,5 TOTAL 6
  Composition of an envelope of formula B:
  Formula B Composition (g) Pectin 1 B-glucan oatmeal 0.25 High-grade polymerization inulin 1 Inulin of low degree of polymerization 0.75 Polydextrose 2.5 Guar gum partially hydrolyzed 0,5 TOTAL 6
  Arms: A: 1 dosis
Dietary Supplement: B: 2 dosis — 1 dosis (3E+09 cfu/d + 12 g of fiber) Two different combinations of fibers (formula A and B) will be tested with the following administration pattern for both groups.
  Week 1: Formula A Week 2: Formula A Week 3: Formula B Week 4: Formula B
  Composition of an envelope of formula A:
  Formula A Composition (g) Pectin 1 B-glucan oatmeal 0.25 High-grade polymerization inulin 1.75 Inulin of low degree of polymerization 1,5 Polydextrose 1 Guar gum partially hydrolyzed 0,5 TOTAL 6
  Composition of an envelope of formula B:
  Formula B Composition (g) Pectin 1 B-glucan oatmeal 0.25 High-grade polymerization inulin 1 Inulin of low degree of polymerization 0.75 Polydextrose 2.5 Guar gum partially hydrolyzed 0,5 TOTAL 6
  Arms: B: 2 dosis

SUMMARY:
Ulcerative colitis (UC) is an entity of complex etiology where environmental, genetic and intestinal microflora-related factors trigger and perpetuate a chronic inflammation of the gastrointestinal tract. It is suspected that an alteration in primary intestinal microbial colonization (dysbiosis) could trigger, or at least contribute to, said oversized immune response. The hypothesis is that the administration of a series of fibers, could improve the bacterial diversity and repair the dysbiosis that has been seen in patients affected by ulcerative colitis, improving the clinical evolution of it. The primary objective of the present study is to know the impact on the microbiota of patients with UC in remission derived from the administration of dietary fibers. The RETOS study is a pilot project in which a population of patients with UC is tested for the effect on the composition of the microbiota that would have the administration of various combinations of fibers, in addition to the tolerability and acceptance by the patient. The clinical applicability derived from this intervention would be to improve the diversity of intestinal flora of patients with ulcerative colitis.

DETAILED DESCRIPTION:
The Phase 1 study is a pilot project in which a population of patients with UC is tested for the effect on the composition of the microbiota that would have the administration of various combinations of fibers, in addition to the tolerability and acceptance by the patient. The study will include two groups of 20 patients each. One of the groups will receive 6 grams of fiber a day in a single shot with the main meal (group 1) and the other group will receive 12 grams of fiber a day divided into two meals with the main meals (group 2). Two different combinations of fibers (formula A and B) will be tested with the following administration pattern for both groups.

Description of the administration pattern Week 1: Formula A Week 2: Formula A Week 3: Formula B Week 4: Formula B

A second sequential cycle similar to the first one (4 weeks with the same administration pattern) will be repeated in order to confirm the reproducibility of the findings.

The two formulas contain fibers known and commonly used in human nutrition, which were previously tested in in vitro models with human faeces and their ability to promote the growth of butyrate-producing bacterial species that are deficient in patients with colitis was proven ulcerative (Faecalibacterium prausnitzii and Roseburia hominis). The fibers are presented in aluminum envelopes to dissolve in a glass of water, juice, infusion or cold cream (max 37 ° C).

In addition, formulas A and B for group 1 (a single intake per day) include the mixture of probiotics i3.1 in quantity per envelope of 3e + 9 colony-forming units, which contains: Pediococcus acidilactici CECT 7483, Lactobacillus plantarum CECT 7484 and Lactobacillus plantarum CECT 7485 in a 1: 1: 1 ratio. Formulas A and B for group 2 (two intakes per day) include the probiotic i3.1 in quantity per envelope of 1.5e + 09 colony-forming units.

In the two groups, the first week the patients will receive half of the dose with the aim of facilitating the adaptation in those people who usually do not consume fiber. The usual diet, tolerability and patient satisfaction will be controlled through biweekly predefined questionnaires.

ELIGIBILITY:
Inclusion Criteria:

1. Adult patients (from 18 to 65 years old) diagnosed with ulcerative colitis (not distal), of at least 1 year of evolution of the disease.
2. Patient in clinical remission two months prior to inclusion (Simple Colitis Clinical Activity Index (SCCAI) <4) and fecal calprotectin <150 μg / g.
3. At least one outbreak in the last year that required systemic corticosteroids or escalating treatment (initiation of thiopurines, optimization of thiopurines, initiation of anti-TNF-alpha, intensification of anti-TNF-alpha, initiation of vedolizumab). At the time of entry into the study, the patient must carry with stable medication at least 2 months in the case of anti-TNF-alpha and mesalazine and 5 months in the case of thiopurine, and without treatment with corticosteroids

Exclusion Criteria:

* Patients with ulcerative proctitis only
* Patients who have received antibiotics the month prior to inclusion until completion
* Usual consumption of probiotics excluding fermented milk (yogurt, kefir ...).
* Supplementation with dietary fiber (without taking into account the one administered in the study).
* The smoking habit is allowed, although the beginning or abandonment of it from two months before the end of the study will have to be documented.
* Patients undergoing hypocaloric diets
* Patients with stenosis or intestinal surgery
* Patients with primary sclerosing cholangitis
* Patients under treatment with ursodeoxycholic acid
* Patients under treatment with ion exchange resins
* Patients under treatment with acenocoumarol (Sintrom)
* The taking of proton pump inhibitors (PPIs) is allowed but their consumption must be controlled, not allowing them to start or suspend their intake during the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2018-03-08 (Actual); Primary Completion 2019-07-02 (Actual); Study Completion 2020-07-02 (Actual)

PRIMARY OUTCOMES:
To know the impact on the microbiota diversity by 16S rRNA analysis of patients with UC in remission derived from the administration of a new product based on dietary fibers | 12 weeks
  The phyla and genera relative abundance analysed by 16S rRNA before and after treatment with the two levels of fiber

SECONDARY OUTCOMES:
To study the tolerability of the product through questionnaires | 4 months
  Change from baseline in tolerability scores using the DHRS scale (0 no pain-5 severe pain) every 15 days
To study the satisfaction of the product through questionnaires | 4 months
  Change from baseline in satisfaction scores using a (0 do not like-10 like a lot)scale every 15 days

CONTACTS AND LOCATIONS:
Overall Officials: Ariana Salavert, PhD, Study Director — Ab-biotics
Locations (1):
- Hospital Vall d'Hebron, Barcelona, Spain